CLINICAL TRIAL: NCT03857347
Title: A Feasibility Study for a Psycho-education Intervention for People With a Functional Neurological Disorder.
Brief Title: Psychoeducation Group Intervention for FND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CAHSS189/05; 18/NS/0137 (Other: NHS Grampian Research Ethics Committee 2)
Record Dates: First submitted 2019-01-21; First posted 2019-02-27 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Functional Neurological Disorder
Keywords: FND; Functional Neurological Disorder; Psychoeducation
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Intervention Model Description: Data will be explored using the reliable and clinically significant change analysis (Morely, Williams & Hussain, 2008). This analysis allows pre and post treatment scores to be compared to see if participants have achieved a level of difference that could be categorized as real and not due to measurement error. Furthermore this score can be helpful to determine if the change seen is clinically significant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief Psychoeducation Intervention (Experimental): 2 group session psychoeducation intervention feasibility study
  Interventions: Other: Psychoeducation Group for FND

INTERVENTIONS:
Other: Psychoeducation Group for FND — he intervention is a psychoeducation based group.

SUMMARY:
This study aims to assess the feasibility of running a brief psychoeducation group intervention in an outpatient setting to assess the practicalities and benefits of offering this type of intervention for both clinicians and patients

DETAILED DESCRIPTION:
A Functional Neurological Disorder (FND) is when the brain has difficulties sending and receiving signals . As a result people can experience problems in how their body and senses work, but there is no physical problem to treat.

Currently there is little treatment to offer after diagnosis, this study will investigate the feasibility and potential benefit to offering a group intervention to people with FND. This group intervention will offer chance to access information and the opportunity to meet others with the similar difficulties. Eligible participants will be those currently attending neurology clinics within NHS Grampian. Participants will complete prior to, during and at 3 months after the group is completed. These measures include health care use of participants, reported physical symptoms, subjective quality of ife and mood we will also take a brief measure of attention and concentration. Reported physical symptoms, subjective quality of life and mood will also be collected before the first group and at the last group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18-64 years with a diagnosis of FND

Exclusion Criteria:

* Anyone the clinical neuropsychologist/neurologist feels, as a result of their clinical judgement, lacks capacity to consent.
* People who are unable to understand the information sheet due to English not being their first language.
* Severe sensory impairment.
* Anyone experiencing active severe psychiatric symptoms
* A dependency on alcohol or recreational drugs
* Learning disability as classified by ICD 10.
* Those unable to travel independently to attend group sessions due to the severity of their symptoms

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
The Medical Outcome Study 36-item Short Form Health Survey (SF-36) | Baseline, Change from Baseline at Time 1 (2 weeks prior to group), Change from Baseline at Time 2 (4 weeks after Time 1), Time 3 change from baseline 3 months from Time 2
  This outcome will measure potential change in self-reported health related quality of life using eight subscales

CONTACTS AND LOCATIONS:
Overall Officials: Dr Pauline M Insch, Principal Investigator — University of Edinburgh/NHS Grampian
Locations (1):
- NHS Grampian, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No